CLINICAL TRIAL: NCT00978042
Title: Safety and Effectiveness of Juvéderm® VOLUMA XC Injectable Gel for Cheek Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: VOLUMA-002
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-09

CONDITIONS: Mid-facial Volume Deficit Related to Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- VOLUMA® XC Treatment Arm (Experimental): Participants treated with JUVÉDERM® VOLUMA® XC Injectable Gel, volume determined by the investigator (up to 12 mLs) at study start. Participants were eligible for re-treatment if applicable.
  Interventions: Device: Juvéderm® VOLUMA XC
- Control Arm_No Treatment then VOLUMA® XC (Other): No treatment for 6 months, then participants were treated with JUVÉDERM® VOLUMA® XC Injectable Gel, volume determined by the investigator (up to 12 mLs). Participants were eligible for re-treatment if applicable.
  Interventions: Device: Juvéderm® VOLUMA XC

INTERVENTIONS:
Device: Juvéderm® VOLUMA XC — Treating Investigator determines the appropriate volume of VOLUMA XC to be injected up to a maximum total of 12 mL for initial and touch-up treatment. One repeat treatment with up to 12 mL may be performed at the Subject's option after study completion.

SUMMARY:
Multicenter, single-blind, randomized, "no-treatment" control study to demonstrate the safety and effectiveness of VOLUMA XC for deep injection for cheek augmentation to correct age-related volume deficit in the mid-face.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 35-65 years of age
* Zygomaticomalar region, anteromedial cheek, submalar region, and/or overall mid-facial volume deficit assessed by the Treating Investigator as grade 3, 4, or 5 on the photometric Mid-Face Volume Deficit Scale (MFVDS)
* Desire cheek augmentation to correct age-related volume deficit in the mid-face
* Accept the obligation not to receive any other facial procedures or treatments affecting facial volume deficit at any time during the study

Exclusion Criteria:

* Received (or is planning to receive) anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti-inflammatory drugs [oral/injectable corticosteroids or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)], or other substances known to increase coagulation time from 10 days pre- to 3 days post injection [Study device injections may be delayed as necessary to accommodate this 10-day wash-out period.]
* Have undergone facial plastic surgery (with the exception of rhinoplasty more than 2 years prior to enrollment), tissue grafting, or tissue augmentation with silicone, fat, or other permanent, or semi-permanent dermal fillers or be planning to undergo any of these procedures at any time during the study
* Have undergone temporary facial dermal filler injections with hyaluronic acid-based fillers within 12 months, porcine-based collagen fillers within 24 months, or neuromodulator injections, mesotherapy, or resurfacing within 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study
* Have begun use of any new over-the-counter or prescription, oral or topical, anti-wrinkle products in the treatment area within 90 days prior to enrollment or be planning to begin use of such products at any time during the study.
* Have very thin skin in the mid-facial region, tendency to accumulate fluid in the lower eyelids, or large infraorbital fat pads
* Have mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy, partial lipodystrophy, inherited disease, or HIV-related disease
* Have a history of anaphylaxis, multiple severe allergies, atopy, or allergy to lidocaine (or any amide-based anesthetic), hyaluronic acid products, or Streptococcal protein, or have plans to undergo desensitization therapy during the term of the study
* Have noticeable acne scarring, an active inflammation, infection, cancerous or pre-cancerous lesion, or unhealed wound or have undergone radiation treatment in the area to be treated

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Los Angeles, California, United States
- Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Jones D, Murphy DK. Volumizing hyaluronic acid filler for midface volume deficit: 2-year results from a pivotal single-blind randomized controlled study. Dermatol Surg. 2013 Nov;39(11):1602-12. doi: 10.1111/dsu.12343. Epub 2013 Oct 4. PMID 24093664
- [Derived] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 345 participants were originally recruited for treatment at 15 sites.
Pre-assignment Details: Prior to randomization, 16 patients were excluded as screen failures and the first two participants per site (30 total) were treated as run-in participants. Of the 299 randomized participants, 17 were discontinued prior to treatment, leaving a "modified intent-to-treat" population of 282 participants (235 in Treatment Arm and 47 in Control Arm).
Period: Initial Treatment Period
Arm/Group | VOLUMA® XC Treatment Arm | Control Arm_No Treatment Then VOLUMA® XC
Started | 235 | 47
MITT_treated With VOLUMA XC | 235 | 35
Completed | 174 (Completed 24-month Follow-Up) | 32
Not Completed | 61 | 15
Not completed — Treated in Error | 0 | 3
Not completed — Ineligibility | 1 | 0
Not completed — Lost to Follow-up | 21 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Discontinuation by Investigator/Sponsor | 2 | 0
Not completed — Consent withdrawn | 22 | 9
Not completed — Other Miscellaneous Reasons | 13 | 0
Period: Received Repeat Treatment
Arm/Group | VOLUMA® XC Treatment Arm | Control Arm_No Treatment Then VOLUMA® XC
Started | 141 (Participants who were deemed eligible for re-treatment.) | 26 (Participants who were deemed eligible for re-treatment.)
Completed | 98 (Completed=Completed Repeat Treatment Follow-up) | 23
Not Completed | 43 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VOLUMA® XC Treatment Arm | Control Arm_No Treatment Then VOLUMA® XC | Total
Number analyzed (Participants) | 235 | 47 | 282
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (7.18) | 54.7 (5.95) | 54.4 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 37 | 226
  Male | 46 | 10 | 56
Region of Enrollment [Number; unit: participants]
  United States | 208 | 41 | 249
  Canada | 27 | 6 | 33

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Based on Improvement in Score on Validated 6-point Mid-Face Volume Deficit Scale (MFVDS)
Description: The primary effectiveness variable was responder rate for the treatment group. The investigator evaluated the volume deficit of the patient's face using the MFVDS 6-point scale where: 0=none (best) to 5=severe (worst). To be considered a "responder," the average of the blinded, independent Evaluating Investigators' assessments of the participant's overall score on MFVDS at 6 months had to be improved (reduced) by ≥ 1 grade compared with the average of the Evaluating Investigator pre-treatment assessments.
Time Frame: 6 months
Population: Participants from the Modified-intent-to-treat (MITT) population, all participants randomized to treatment who received treatment and all participants randomized to "no treatment" control arm, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | VOLUMA® XC Treatment Arm | Control Arm_No Treatment Then VOLUMA® XC
Number analyzed (Participants) | 209 | 36
percentage of responders | 85.6 [NA to NA] — Only a 97.5% Confidence Interval was calculated = 79.33% to 90.64%. | 38.9 [NA to NA] — Only a 97.5% Confidence Interval was calculated = 21.33% to 58.82%.

2. Secondary Outcome: Duration of Treatment Effect
Description: Duration of treatment effect was determined by Kaplan-Meier (KM) product limit estimate of the percentage of participants in the treatment group that maintained at least a 1-point improvement in the overall mid-face volume deficit score on the Mid-Face Volume Deficit Scale (MFVDS) based on the average of the 2 blinded Evaluating Investigators' assessments (with 95% Greenwood's Confidence Interval).
Time Frame: 24 Months
Population: Participants from the Modified-intent-to-treat (MITT) population, all participants randomized to the treatment arm who received treatment and all participants randomized to "no treatment" control arm who received treatment, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VOLUMA® XC Treatment Arm | Control Arm_No Treatment Then VOLUMA® XC
Number analyzed (Participants) | 235 | 35
Percentage of participants | 44.6 [37.31 to 51.87] | 44.9 [27.76 to 62.14]

3. Secondary Outcome: Responder Rate Based on Improvement in Score on Global Aesthetic Improvement Scale (GAIS)
Description: The investigator evaluated the patient's overall mid-face volume using the GAIS 5-point scale where: 2=much improved to -2=much worse. To be considered a "responder," the average of the blinded, independent Evaluating Investigators' assessments of the participant's overall score on GAIS at 6 months had to be improved (reduced) by ≥ 1 grade compared with the average of the Evaluating Investigator pre-treatment assessments.
Time Frame: 6 months
Population: Only those participants from the Modified-intent-to-treat (MITT) population randomized to the Treatment Arm who received treatment with available data are included in the analysis.
Measure: Number; unit: Percentage of responders
Arm/Group | VOLUMA® XC Treatment Arm
Number analyzed (Participants) | 209
Percentage of responders | 81.8 [NA to NA]

4. Secondary Outcome: Responder Rate Based on Improvement in Score on MFVDS by Facial Region
Description: The investigator evaluated the volume deficit of the patient's face using the MFVDS 6-point scale where: 0=none (best) to 5=severe (worst). To be considered a "responder," the average of the blinded, independent Evaluating Investigators' assessments of the participant's respective mid-facial area score on MFVDS at 6 months had to be improved (reduced) by ≥ 1 grade compared with the average of the Evaluating Investigator pre-treatment assessments. The percentage of responders is categorized by facial region.
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of responders
Arm/Group | VOLUMA® XC Treatment Arm
Number analyzed (Participants) | 209
percentage of responders
  Zygomaticomalar Region | 75.6 [NA to NA]
  Anteromedial Cheek | 83.3
  Submalar Region | 77.0

ADVERSE EVENTS:
Time Frame: 30 days after repeat treatment (Up to 28 months)
Description: Only device- or procedure-related Serious Adverse Events (SAEs) are reported. All Adverse Events (AEs) occurring at >5% frequency are reported. More than 1 event can occur in 1 participant.
Groups:
- All Treated Participants_ AEs Initial Treatment: All participants in the original VOLUMA® XC Treatment Arm and all participants in the No Treatment then VOLUMA® XC Arm (who received delayed treatment) treated with JUVÉDERM® VOLUMA® XC Injectable Gel, volume determined by the investigator (up to 12 mLs). AEs reported are AEs with onset prior to retreatment.
- All Treated Participants_ AEs After Repeat Treatment: All participants in the original VOLUMA® XC Treatment Arm and all participants in the No Treatment then VOLUMA® XC Arm (who received delayed treatment) treated with JUVÉDERM® VOLUMA® XC Injectable Gel, volume determined by the investigator (up to 12 mLs) and who received re-treatment. AEs reported are AEs with onset after retreatment.
Arm/Group | All Treated Participants_ AEs Initial Treatment | All Treated Participants_ AEs After Repeat Treatment
Serious Adverse Events (participants affected / at risk) | 11/270 | 2/167
Other Adverse Events (participants affected / at risk) | 98/270 | 15/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Participants_ AEs Initial Treatment (N=270) | All Treated Participants_ AEs After Repeat Treatment (N=167)
Inflammation (General disorders) | 1 | 0
Injection site mass (General disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Optic neuropathy (Eye disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants_ AEs Initial Treatment (N=270) | All Treated Participants_ AEs After Repeat Treatment (N=167)
Injection site mass (General disorders) | 54 | 8 — Administration site condition
Injection site induration (General disorders) | 39 | 7 — Administration site condition
Injection site swelling (General disorders) | 21 | 1 — Administration site condition
Injection site pain (General disorders) | 17 | 1 — Administration site condition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with Allergan.